CLINICAL TRIAL: NCT02335164
Title: A Randomised, Controlled, Blinded Phase 1 Study to Evaluate the Immunogenicity and Safety of a Pandemic Avian H5 Influenza Vaccine in Adults
Brief Title: A Phase 1 Study to Evaluate the Immunogenicity and Safety of a Pandemic Avian Influenza Vaccine in Adults
Acronym: FLU003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Flinders University (Other); Australian Respiratory and Sleep Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FLU003
Record Dates: First submitted 2015-01-04; First posted 2015-01-09 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- HA 45ug (Experimental): recombinant influenza hemagglutinin (H5) 45ug, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin
- HA 45ug+Advax1 (Experimental): recombinant influenza hemagglutinin(H5) 45ug, Advax1 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax1
- HA 45ug+Advax2 (Experimental): recombinant influenza hemagglutinin (H5) 45ug, Advax2 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax2
- HA 15ug+Advax1 (Experimental): recombinant influenza hemagglutinin (H5) 15ug, Advax1 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax1
- HA 15ug+Advax2 (Experimental): recombinant influenza hemagglutinin (H5) 15ug, Advax2 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax2
- HA 5ug+Advax1 (Experimental): recombinant influenza hemagglutinin (H5) 5ug, Advax1 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax1
- HA 5ug+Advax2 (Experimental): recombinant influenza hemagglutinin (H5) 5ug, Advax2 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax2
- HA 2.5ug+Advax2 (Experimental): recombinant influenza hemagglutinin (H5) 2.5ug, Advax2 adjuvant 20mg, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin; Biological: Advax2
- HA 15ug (Experimental): recombinant influenza hemagglutinin (H5) 15ug, i.m. injection, 2 doses
  Interventions: Biological: recombinant influenza hemagglutinin

INTERVENTIONS:
Biological: recombinant influenza hemagglutinin — recombinant influenza hemagglutinin
Biological: Advax1 — Delta inulin adjuvant formulation 1
  Arms: HA 15ug+Advax1; HA 45ug+Advax1; HA 5ug+Advax1
Biological: Advax2 — Delta inulin adjuvant formulation 2
  Arms: HA 15ug+Advax2; HA 2.5ug+Advax2; HA 45ug+Advax2; HA 5ug+Advax2

SUMMARY:
Recombinant hemagglutinin has been shown to induce protective neutralising antibodies against avian influenza virus but is relatively non-immunogenic. An ideal pandemic avian influenza influenza vaccine would combine hemagglutinin antigen with an appropriate adjuvant to increase its immunogenicity. This Phase 1 study will collect preliminary human safety and efficacy data on combined formulations of recombinant hemagglutinin with Advax adjuvant formulations administered by intramuscular injection

DETAILED DESCRIPTION:
This is a study to test new vaccine formulations against pandemic avian influenza ("bird flu"). Bird flu is a potentially deadly disease that is caused by influenza virus from birds. It is not the same as the common seasonal flu for which there is a seasonal vaccine released around March each year. To date, bird flu due to the H5N1 strain of influenza virus has infected over 500 people mainly in Asia resulting in death in more than half the cases. More recently there has been an outbreak of another bird flu virus in China known as H9N7 that is also highly lethal when it infects humans. Vaccination is the single most effective measure to prevent infection from bird flu viruses such as H5N1 or H9N7 should such a pandemic occur. In the event of a major bird flu pandemic outbreak, vaccine supplies are likely to be very limited, as there is not currently sufficient manufacturing capacity to provide enough vaccine quickly for the whole population. Research is needed on how to make the pandemic flu vaccine more effective but also how to stretch vaccine supplies using a strategy called 'antigen-sparing'. This can potentially be achieved by using an important ingredient called an 'adjuvant'. Adjuvants act by stimulating the immune system to make vaccines more effective. This study will test Advax adjuvants which are based on delta inulin in combination with recombinant hemagglutinin from the H5N1 influenza virus serotype.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory males or females aged 18 years and over
* Able to provide written informed consent
* Willing and able to comply with the protocol for the duration of the study.
* Not planning to have seasonal influenza vaccine within 2 months from the time of the first trial immunization

Exclusion Criteria:

* Pregnant or lactating women.
* Women of childbearing potential unless using a reliable and appropriate contraceptive method.
* Receipt of another investigational agent within 28 days preceding initiation of treatment.
* Any other serious medical, social or mental condition which, in the opinion of the investigator, would be detrimental to the subjects or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events | 12 months
  The frequency of adverse events will be compared between groups

SECONDARY OUTCOMES:
Hemagglutination inhibition assay | 1 month post each immunization and 11 months post final immunization
  Seroconversion, seroprotection and GMT fold increase will be compared between groups at each time point using hemagglutination inhibition titers

OTHER OUTCOMES:
Plasmablast response | 7 and 28 days post each immunization
  The size of the plasmablast response will be compared between groups as an experimental endpoint
T-cell response | 7 and 28 days post each immunization
  The size of the memory T cell response will be compared between groups as an experimental endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, FRACP, PhD, Principal Investigator — Flinders University
Locations (1):
- Flinders University, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided